CLINICAL TRIAL: NCT02068742
Title: Postoperative Cognitive Dysfunction in Elderly
Acronym: ElderlyPOCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Paolo Severgnini, MD, PhD, Università degli Studi dell'Insubria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1048
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: post-operative cognitive dysfunction; elderly; Mini Mental State Examination; Geriatric Index of Comorbidity; Geriatric Depression Scale; Trail Making Test B-A; Digit Span; Digit Symbol Substitution Test
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: First arm of the study considers patients from the operating room with general anesthesia; Second arm of the study considers patients from geriatric regular general ward, without any anesthesia.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Anesthesia patients battery neuropsychological tests (Experimental): Mini Mental State Examination, Geriatric Index of Comorbidity, Geriatric Depression Scale, Trail Making Test B-A, Digit Span, Digit Symbol Substitution Test Application of the scores will be on the day 0 (the day before the surgery), day 2 and day 4 (after the surgery).
  Interventions: Other: battery neuropsychological tests
- Regular recovery patients (Active Comparator): Mini Mental State Examination, Geriatric Index of Comorbidity, Geriatric Depression Scale, Trail Making Test B-A, Digit Span, Digit Symbol Substitution Test Application of the scores will be on the day 0 (the day after the hospital admission), day 2 and day 4 (days after the hospital admission).
  Interventions: Other: battery neuropsychological tests

INTERVENTIONS:
Other: battery neuropsychological tests — Application of the scores will be on the day 0 (the day before the surgery), day 2 and day 4 (after the surgery).
  Other Names: Mini Mental State Examination,; Geriatric Index of Comorbidity,; Geriatric Depression Scale,; Trail Making Test B-A,; Digit Span,; Digit Symbol Substitution Test

SUMMARY:
Interventional Study of Early Postoperative Cognitive Dysfunction in Elderly Patients Undergoing General Anesthesia

The main purpose of this study is to determine the incidence of early postoperative cognitive dysfunction in elderly patients and its time course.

This study will first evaluate the preoperative cognitive function of elderly patients based on several criteria including complete patient history, laboratory and instrumental exams, and the following measures in order to identify conditions and pathologies that may influence cognitive function.

* Mini Mental State Examination
* Geriatric Index of Comorbidity
* Geriatric Depression Scale

The following neuropsychological tests will be performed on the same day within 7 days of surgery (baseline):

* Trail Making Test B-A
* Digit Span
* Digit Symbol Substitution Test

The three cognitive function assessments will be repeated at the following postoperative time points and the change from the preoperative baseline to each time will be evaluated:

* Day 2 (time point 1)
* Day 4 (time point 2)
* Between days 85 and 90 (time point 3)

If the patient seems confused before the postoperative administration of these tests, the Neecham Confusion Scale will be used to evaluate the patient for the presence of postoperative delirium; if delirium is not detected, the cognitive function tests will be administered.

DETAILED DESCRIPTION:
This study has three specific aims:

1. To define the frequency of occurrence of early post-operative cognitive dysfunction and its time course.
2. To assess risk factors for the onset of post-operative cognitive dysfunction and possible causal factors.
3. to compare our results with those from the international literature.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Surgery scheduled under general anesthesia, that is expected to last 90 minutes or longer for the arm experimental

Exclusion Criteria:

* A score of 20 or less on the Mini-Mental State Examination (MMSE)
* Illiteracy
* Can't understand Italian language
* Serious hearing or vision impairment not treatable
* A history of any disease of the central nervous system
* A current or past history of psychiatric illness
* A current use of major tranquilizers or antidepressants
* alcoholism or drug dependence or abuse
* Scheduled to undergo cardiac, carotid or intracranial procedures
* Not expected to be alive or available to complete testing at 90 days after surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
frequency of occurrence of post-operative cognitive dysfunction | about 90 days
  we apply specific neuropsychological tests find out post-operative cognitive dysfunction in elderly patients (number of patients 80)

SECONDARY OUTCOMES:
assess risk factors and causal factors in the onset of post-operative cognitive dysfunction (number of patients 80) | about 90 days
  we look for possible risk factors or causal factors in the onset of post-operative cognitive dysfunction considering comorbidity of patients and specific events occurred during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Severgnini Paolo, MD, PhD, Study Director — Università degli Studi dell'Insubria
Locations (1):
- Ospedale di Circolo e Fondazione Macchi, Varese, Italy